CLINICAL TRIAL: NCT00575679
Title: Behavior and Driving Safety Study
Acronym: BADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Sacramento Police Department (Unknown); California Office of Traffic Safety (Other Government); University of Michigan (Other); Robert Wood Johnson Foundation (Other); Teachable Moment Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 243197; UCDIRB-200614967; OTS-AL0757 (Other: UC Davis)
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Alcoholic Intoxication
Keywords: Automobile driving; Driving under the influence; Interview, psychological; Brief intervention; Brief motivational interview
MeSH Terms: conditions — Alcoholic Intoxication; Driving Under the Influence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Brief motivational interview
  Interventions: Behavioral: Brief motivational interview
- 2 (No Intervention): No discussion

INTERVENTIONS:
Behavioral: Brief motivational interview — The brief motivational interview is a non-confrontational, patient-centered discussion between a counselor (e.g., social worker, nurse, physician, or psychologist) and an at-risk individual during which the individual's motivation and confidence to change health-related behaviors are explored.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether brief motivational interviews reduce the likelihood of driving under the influence of alcohol (DUI).

DETAILED DESCRIPTION:
Despite extensive legislative, law enforcement, and public awareness efforts, driving under the influence of alcohol (DUI) remains a major cause of mortality and loss of years of productive life. A brief motivational interview (BI) is a non-confrontational, patient-centered discussion during which the individual's motivation and confidence to change health-related behaviors are explored. Previous studies of BIs in health care settings suggest that BIs administered after hospitalization for alcohol-related injury reduce the likelihood of repeat injury hospitalization and arrest for DUI.

ELIGIBILITY:
Inclusion Criteria:

* Second or greater arrest for driving under the influence of alcohol
* Arrest involved operation of a motor vehicle
* At least 18 years of age
* English-speaking

Exclusion Criteria:

* Arrest involved injury to another person
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

PRIMARY OUTCOMES:
Time to repeat arrest for driving under the influence of alcohol | Up until one year after the conclusion of enrollment

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test score | 6 and 12 months
Time to alcohol-related injury hospitalization | Up until one year after the conclusion of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Garth H Utter, MD MSc, Principal Investigator — University of California, Davis; Leon J Owens, MD, Study Director — University of California, Davis
Locations (1):
- Sacramento County Main Jail, Sacramento, California, United States